CLINICAL TRIAL: NCT02567851
Title: BREVITY: A Phase II Study of Brentuximab Vedotin Using a Response Adapted Design in Patients With Hodgkin Lymphoma Unsuitable for Chemotherapy Due to Age, Frailty or Co-morbidity
Brief Title: A Study of Brentuximab Vedotin in Patients With Hodgkin Lymphoma Unsuitable for Chemotherapy Due to Age, Frailty or Co-morbidity
Acronym: BREVITY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Leukaemia Lymphoma Research (Other); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG_11-225; 2012-000214-11 (EudraCT Number)
Record Dates: First submitted 2015-09-29; First posted 2015-10-05 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2017-11

CONDITIONS: Hodgkin Disease
Keywords: Brentuximab Vedotin; PET scans; Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brentuximab Vedotin (Experimental): brentuximab vedotin will be administered at an initial dose of 1.8 mg/kg every 3 weeks as a 30-minute outpatient i.v. infusion. A maximum of 16 cycles
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — Monoclonal antibody drug conjugate
  Other Names: Adcetris

SUMMARY:
An early phase II, single arm, two stage study, to investigate the level of activity, duration of response and tolerability of brentuximab vedotin (SGN-35), as a single agent, utilising a response adapted approach, in older, frailer or co-morbid patients with previously untreated Hodgkin lymphoma.

Opened Feb 2014 and will recruit over 18 months. Duration of treatment will be dependent on the patients' response (see schema below) with a maximum of 16 cycles over 48 weeks.

At the end of treatment patients will be assessed clinically at 3 months intervals and by CT scan at 15, 18, 24 and 36 months. For those still alive and disease free after 2 years, follow-up will be according to local practice.

DETAILED DESCRIPTION:
Stage 1 will recruit 20 patients. If at least patients 8 respond after the initial 4 cycles of SGN-35 a further 10 patients will be recruited to stage 2.

In all cases brentuximab vedotin will be administered at an initial dose of 1.8 mg/kg every 3 weeks as a 30-minute outpatient i.v. infusion.

After baseline staging (including PET and CT scans (PET0 + CT0), performed on PET scanners approved for the purpose by The PET Imaging Centre at St Thomas'/Guy's), all eligible and consenting patients will receive an initial 4 cycles of brentuximab vedotin following which response and continuation of brentuximab vedotin will be assessed by PET (PET4) in the first instance. Patients achieving CMR (Deauville score 1-3) will continue treatment. Patients achieving PMR (Deauville score 4,5 with uptake less than baseline) will also continue treatment. Patients achieving NMR (Deauville score 4,5 with no change in uptake from baseline) or PMD (Deauville score 4,5 with increased intensity of uptake compared to baseline and/or new lesions consistent with lymphoma) will stop brentuximab vedotin and be considered for alternative therapy.

CT4 will be performed for future comparison with CT8, CT12 and CT 16 (to exclude Progressive Disease (PD) and to correlate metabolic and radiological responses) and to inform continued treatment. Patients not achieving Deauville score 1-3 at PET 4 will also have a PET scan at completion of treatment (after 16 cycles or earlier if brentuximab vedotin discontinued for reasons other than PD)

In addition an exploratory PET scan will be performed after 2 cycles of brentuximab vedotin (PET2); investigators will be blinded to the results of PET2 which will not influence patient management in any way. All PET scans will be centrally reviewed for QA purposes by The PET Imaging Centre at St Thomas'/Guy's, under the supervision of Sally Barrington and Mike O'Doherty, using the framework developed for the recently completed RAPID and RATHL trials. CT scans after 4 cycles and at the end of treatment may also be reviewed.

After the initial 4 cycles of brentuximab vedotin, subsequent treatment will be response adapted according to PET scan result the following schedule:

* Those with a Complete Metabolic Response (CMR, Deauville Score 1, 2 or 3) at PET 4 will receive up to 12 additional cycles of brentuximab vedotin (maximum of 16 cycles) depending on no evidence of PD by a CT scan performed after each group of 4 cycles of brentuximab vedotin.
* Patients with a Partial Metabolic Response (PMR) at PET4 will receive up to 12 additional cycles of brentuximab vedotin (maximum of 16 cycles) depending on no evidence of PD on a CT scan performed after each group of 4 cycles of brentuximab vedotin.
* Patients with No Metabolic Response (NMR) will stop brentuximab vedotin and be considered for alternative therapy.
* Patients with progressive disease at any time as determined by either CT or PET scan performed after each group of 4 cycles of brentuximab vedotin or in response to clinical concerns will stop study treatment and receive subsequent therapy at investigator discretion. Clinical concerns over PD should be confirmed by either a CT or PET scan.
* Patients who come off treatment with brentuximab vedotin for any other reason (toxicity, patient decision, investigator advice) should have a CT scan performed for response assessment. In addition patients with Partial Metabolic Response at PET 4 should also have a PET scan performed.

All patients who have not progressed irrespective of how many cycles of brentuximab vedotin received will be clinically assessed every 3 months and have a CT scan at months 3, 6, 9, 12. These scan may take place during therapy. During follow-up CT scans will be performed 15, 18, 24 and 36 months from the start of treatment. For those still alive and disease-free after 3 years following start of treatment, follow-up will be according to local practice but data recorded must include date of progressive disease, type of any subsequent therapies, date and cause of death.

For patients who progress at any time, follow-up will be according to local practice but data must be recorded for 5 years form the start of treatment and must include date of progressive disease, type of any subsequent therapies, date and cause of death.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed CD30 positive classical Hodgkin lymphoma
2. No previous treatment for classical Hodgkin lymphoma
3. Aged ≥ 16 years
4. Stages II (with B symptoms, extranodal disease, bulky disease, ≥3 sites of nodal involvement, fewer than 3 sites of nodal involvement but unsuitable for radiotherapy because of anatomical distribution or ESR ≥50 mm/h), III and IV classical Hodgkin lymphoma
5. Any of the following:

   At any age and with ECOG score of 0, 1, 2 or 3, for whom standard chemotherapy considered inappropriate because:
   * Impaired cardiac function defined either by an ejection fraction of < 50% assessed by echocardiogram or nuclear medicine scan (MUGA)
   * Left ventricular ejection fraction ≥50% measured by echocardiography or MUGA but in the presence of significant co-morbidities or cardiac risk factors such as diabetes mellitus, hypertension, peripheral vascular disease, ischaemic heart disease, previous myocardial infarction, obesity, stroke or transient ischaemic attacks (TIA) that make anthracycline-containing chemotherapy inadvisable as determined by the investigator.
   * Heart failure clinically determined by the presence of New York Heart Association (NYHA) heart failure grade II and III due to a cause other than Hodgkin Lymphoma
   * Impaired respiratory function with DLCO and/or FVC/FEV1 ratio <75% of predicted due to a cause other than Hodgkin lymphoma

   For patients aged 60 years or older,
   * an ECOG score of 1, 2 or 3 for any reason, before the start of permitted steroids (see section 7.9) and considered unsuitable for treatment with standard chemotherapy by the investigator

   All co-morbidities must be documented on the baseline form and the CIRS-G score (if 60 years or older) recorded.
6. FDG avid disease - proven by PET scan
7. Measurable disease with at least one lesion measuring >1.5 cm in long axis diameter (for nodal lesions) or >1.0cm in long axis diameter (for extra-nodal lesions)
8. Written informed consent
9. Able to comply with requirements of the protocol (including PET scans)
10. Agree and be able to use adequate contraception if required

Exclusion Criteria:

1. Nodular lymphocyte predominant Hodgkin lymphoma
2. Grade 2 or worse peripheral neuropathy
3. Haemoglobin <90 g/L (transfusion allowed)
4. Unsupported neutrophil count <1.0 x 109/l and platelet count <100 x 109/l unless due to bone marrow infiltration by Hodgkin lymphoma demonstrated by trephine biopsy
5. Serum bilirubin ≥1.5 times upper limit normal unless due to Hodgkin lymphoma or Gilbert's syndrome
6. Creatinine clearance <30 ml/min (calculated by the modified Cockroft-Gault formula, see appendix) unless due to Hodgkin lymphoma. Patients with an eGFR <30 ml/min but a measured GFR by another method (e.g. EDTA) of 30ml/min or greater would be eligible.
7. Pregnant or lactating women
8. Any other cancer diagnosis within the last 24 months - except for:

   * Appropriately treated superficial melanoma, basal cell carcinoma and squamous cell carcinoma of the skin
   * Appropriately treated cervical intra-epithelial neoplasia
   * In situ or organ confined prostate cancer not currently requiring therapy

   Previous cancers treated with curative intent and with no evidence of recurrence following a minimum of at least 2 years of follow-up are permitted.
9. The use of other investigational or anti-neoplastic agents within the previous 6 weeks or during the trial.
10. Known to be HIV, Hep B positive (Hep B Core antibody positive allows inclusion providing surface / core antigen both negative) or Hep C positive (Hep C antibody positive allows inclusion providing PCR for viral RNA is negative).
11. Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin.
12. Known cerebral or meningeal involvement by Hodgkin lymphoma
13. Symptoms or signs of progressive multifocal leukoencephalopathy (PML)
14. Any active systemic viral, bacterial, or fungal infection requiring intravenous antimicrobials within 2 weeks prior to registration
15. Evidence of current uncontrolled cardiovascular conditions, including unstable angina and NYHA grade IV heart failure
16. ECOG 4 at registration

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01-14 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Complete metabolic response rate (CMR) after 4 cycles of brentuximab vedotin defined as Deauville score of 1, 2 or 3 by PET | 4 cycles (3 months)
  The number of patients achieving a CR at PET4 (after cycle 4) with confidence intervals (CIs) will be presented and assessed using the Simons 2-stage design criterion.

SECONDARY OUTCOMES:
Tolerability is defined in terms of absence of toxicities related to BV quantified by the CTCAE v4 criteria and dose intensity. | 16 cycles (1 year from start of treatment)
  Numbers of patients in each CTCAE toxicity category will be reported. Dose intensity will be reported as the median dose intensity together with full range. The number of patients with dose interruptions, dose reductions and number discontinuing treatment will also be reported over the treatment period.
Overall objective response rate (ORR), including complete or partial metabolic response (CMR/PMR), after 4 cycles and 16 cycles of treatment with BV according to The Lugano Classification | 16 cycles (1 year from start of treatment)
  ORR based on the Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification will be presented as the number of patients in each response category (CR/PR), as well as overall.
Progression Free Survival (PFS) where progression is defined as the time from date of Cycle 1 Day 1 until documented progressive disease or death from any cause | 5 years from start of treatment
  Survival estimates (PFS) will be calculated using the Kaplan-Meier method. Median, 12, 24 and 60 month estimates will be presented with CIs. Causes of death will also be reported.
Overall survival (OS) and cause of death. OS is defined as the time from Cycle 1 Day 1 to the date of death from any cause. Alive patients will be censored at their date of last follow-up | 5 years from start of treatment
  Survival estimates (OS) will be calculated using the Kaplan-Meier method. Median, 12, 24 and 60 month estimates will be presented with CIs. Causes of death will also be reported.
Deauville score after cycle 2 based on blinded PET2 scan | 5 years from start of treatment
  Deauville score after cycle 2 (blinded PET2) will be reported as the number of patients in each score category. Scores will also be categorised into complete response (DS=1, 2 or 3) or not complete response (DS=4,5) and reported as the number and proportion of patients in each category
Correlation of Deauville score after 2 cycles (blinded PET2) with Deauville score after 4 cycles (PET 4) | 5 years from start of treatment
  Correlation coefficients will be reported to assess the association of DS after 2 cycles (at blinded PET2) with DS after 4 cycles (at PET 4) will be assessed by cox-regression modelling
Correlation of Deauville score after 2 cycles (blinded PET2) with response after 16 cycles | 5 years from start of treatment
  Correlation coefficients will be reported to assess the association of DS after 2 cycles (at blinded PET2) with end of treatment response. The relationship will also be assessed by cox-regression modelling
Correlation of Deauville score after 2 cycles (blinded PET2) with overall survival | 5 years from start of treatment
  Correlation coefficients will be reported to assess the association of DS after 2 cycles (at blinded PET2) with OS and also will be assessed by cox-regression modelling
Correlation of Deauville score after 2 cycles (blinded PET2) with progression-free survival | 5 years from start of treatment
  Correlation coefficients will be reported to assess the association of DS after 2 cycles (at blinded PET2) with PFS and assessed by cox-regression modelling
CIRS-G profile in the study population assessed at baseline | 5 years from start of treatment
  Numbers of patients in each CIRS-G score at baseline will be reported.
Co-morbidities satisfying eligibility criteria in the study population and documented throughout the study | 5 years from start of treatment
  Numbers of patients will be presented for common co-morbidities (ECOG and IPS) and any additional treatments administered following treatment with brentuximab vedotin

OTHER OUTCOMES:
Differences in Progression Free Survival between patients who continue treatment following PET4 due to CMR and those who continue treatment following PMR at PET4. | 5 years from start of treatment
  Where appropriate secondary outcomes analysis will be repeated to explore differences between patients who continue treatment following PET4 due to CMR and those who continue treatment following PMR at PET4.
Differences in Overall Survival between patients who continue treatment following PET4 due to CMR and those who continue treatment following PMR at PET4. | 5 years from start of treatment
  Where appropriate secondary outcomes analysis will be repeated to explore differences between patients who continue treatment following PET4 due to CMR and those who continue treatment following PMR at PET4.

CONTACTS AND LOCATIONS:
Locations (12):
- United Kingdom (12):
  - Queen Elizabeth Hospital, Birmingham
  - University Hospital of Wales, Cardiff
  - Beatson West of Scotland Cancer Center, Glasgow
  - St James University Hospital, Leeds
  - University Hospital, Leicester
  - Royal Liverpool Hospital, Liverpool
  - Guys Hospital, London
  - The Christie Hospital, Manchester
  - The Freeman Hospital, Newcastle
  - Norfolk and Norwich Hospital, Norwich
  - The Churchill Hospital, Oxford
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Gibb A, Pirrie SJ, Linton K, Warbey V, Paterson K, Davies AJ, Collins GP, Menne T, McKay P, Fields PA, Miall FM, Nagy E, Wheatley K, Reed R, Baricevic-Jones I, Barrington S, Radford J. Results of a UK National Cancer Research Institute Phase II study of brentuximab vedotin using a response-adapted design in the first-line treatment of patients with classical Hodgkin lymphoma unsuitable for chemotherapy due to age, frailty or comorbidity (BREVITY). Br J Haematol. 2021 Apr;193(1):63-71. doi: 10.1111/bjh.17073. Epub 2020 Sep 14. PMID 32926420